CLINICAL TRIAL: NCT04801485
Title: D-chiro Inositol in Prevention of Gestational Diabetes Mellitus in High Risk Pregnant Women in China
Brief Title: D-chiro Inositol in Prevention of Gestational Diabetes Mellitus in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Quzhou Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-20190035-R
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The random number table is compiled by the investigator who is specially responsible for grouping and saved. The investigator packaged and coded drugs according to random number table, and recorded. The packaged and numbered drugs are stored in the enrollment office.
  When the participants meet the inclusion criteria by care providers (doctors), the enrollment office generates a random number for each subject. The participants received the package of drugs according to their random number, and the random number was recorded in the record book.
  If there are adverse events or the subjects request to withdraw from the trial, the investigator should uncover the blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-chiro inositol (Active Comparator): 500 mg twice a day
  Interventions: Dietary Supplement: D-chiro inositol
- Placebo (Placebo Comparator): 500 mg twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-chiro inositol — Active group receives inositol 1 gram per day as well as health guidance about diet and exercise. From recruitment until OGTT.
  Arms: D-chiro inositol
Dietary Supplement: Placebo — Placebo (similar appearance but not containing myo-inositol) 1 gram per day before meals. Similar health guidance about diet and exercise. From recruitment until OGTT.
  Arms: Placebo

SUMMARY:
Inositol is a type of food additives, which plays an important role in insulin signal pathway and is related to insulin sensitivity. Our randomized, double-centered, placebo-controlled study is planned to recruit 360 pregnant women who is in high risk for gestational diabetes. They will be assumed randomly 1 g of D-chiro inositol per day or placebo from 12-16th gestational weeks until Oral Glucose Tolerance Test (OGTT) at 24-28th gestational weeks. Perinatal outcomes about delivery time, neonatal weight will be registered.

ELIGIBILITY:
Inclusion Criteria:

* During 12-16 weeks gestation
* Meet any of the following: prepregnancy BMI > 24, family history of diabetes (type 1 or 2), GDM history, history of delivering macrosomia, gestational history of stillbirth;
* Willing to participate

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus diagnosed before pregnancy
* Multiple gestation
* Mental or cognitive impairment cannot complete the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
the incidence of gestational diabetes | 24-28th weeks gestation
  The number of cases and incidence of gestational diabetes according to OGTT

SECONDARY OUTCOMES:
the perinatal outcomes-1 | Delivery
  the incidence of macrosomia (macrosomia refers to a newborn weighs more than 4 kg)
the perinatal outcomes-2 | Delivery
  weight gain during pregnancy (kg)
the perinatal outcomes-3 | Delivery
  the Caesarean-section incidence (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Xinning Chen, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Chen X, Du Z, Zhang Z, Chen D. D-Chiro Inositol Supplementation and the Occurrence of Gestational Diabetes: A Randomized Controlled Trial in China. Food Sci Nutr. 2024 Dec 5;13(1):e4601. doi: 10.1002/fsn3.4601. eCollection 2025 Jan. PMID 39803251

DOCUMENTS (1):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04801485/Prot_000.pdf